CLINICAL TRIAL: NCT06648265
Title: IMPACT OF TRANEXAMIC ACID IN TUMESCENT SOLUTION ON POSTOPERATIVE OUTCOMES AFTER LIPOSUCTION: A DOUBLE-BLIND, CONTRALATERAL ARM RANDOMIZED CLINICAL TRIAL
Brief Title: EFFECTS OF TRANEXAMIC ACID IN TUMESCENT SOLUTION FOR LIPOSUCTION PROCEDURES
Acronym: ARMTXA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Total Definer Research Group (Other)
Responsible Party: Principal Investigator, Alfredo Hoyos, Plastic Surgeon, Total Definer Research Group
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: ArmsTXA001
Record Dates: First submitted 2024-09-11; First posted 2024-10-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Liposuction; Bruising; Inflammation; Skin Condition; Edema Arm; Ecchymosis; Hematoma
Keywords: Tranexamic Acid; Body contouring; Liposuction; Liposculpture; Patient outcomes; High Definition Liposculpture
MeSH Terms: conditions — Contusions; Inflammation; Skin Diseases; Ecchymosis; Hematoma | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Intervention Model Description: Crossover assignment (each subject serves as their own control with one arm receiving TXA and the other not)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TXA Group (Experimental): Tumescent solution with TXA
  Interventions: Drug: Tranexamic Acid (Topical); Drug: Tumescent solution with dilute lidocaine and epinephrine
- Control Group (Placebo Comparator): Tumescent Solution without TXA
  Interventions: Drug: Tumescent solution with dilute lidocaine and epinephrine

INTERVENTIONS:
Drug: Tranexamic Acid (Topical) — Add 250 mg of TXA per liter of Klein's Tumescent solution for arm liposculpture
  Arms: TXA Group
Drug: Tumescent solution with dilute lidocaine and epinephrine — Arm infiltration with traditional Klein's tumescent solution

SUMMARY:
The goal of this trial is to evaluate the effect of adding Tranexamic Acid (TXA) to the tumescent solution used in arm liposuction on postoperative outcomes. Study population includes healthy volunteer adults undergoing Liposculpture procedures. The main question it aims to answer is:

1. Does Tranexamic acid exert benefit on postoperative outcomes after liposuction? Researchers will compare TXA versus traditional tumescent solution to see if there are benefits on adding it to the tumescent solution.

Participants will undergo High Definition Liposculpture involving arms, legs and their torso. One arm will be infiltrated with traditional Klein's tumescent solution and the other one with the same one but adding Tranexamic Acid.

DETAILED DESCRIPTION:
Study Design:

Allocation: Randomized (one arm with TXA, one without) Intervention Model: Crossover assignment (each subject serves as their own control with one arm receiving TXA and the other not) Masking: Double-blind (Participant and Outcomes Assessor)

Interventions:

Experimental Arm (TXA): Infiltration with Klein's tumescent solution (1000 ml of Ringer's Lactate + Epinephrine 1 mg + Lidocaine 1 mg) plus 250 mg of tranexamic acid.

Control Arm: Infiltration with Klein's tumescent solution (1000 ml of Ringer's Lactate + Epinephrine 1 mg + Lidocaine 1 mg) without tranexamic acid.

Recruitment Information:

Adults aged 18-60 undergoing elective High Definition liposuction. No known allergies to TXA or lidocaine. BMI of 30 kg/m^2.

Study Start Date: January 2022. Primary Completion Date: January 2024. Study Completion Date: June 2024. Study Locations: Clinica Dhara, Bogota DC, Colombia.

Data Collection: Photomicrographic analysis with ImageJ (Fiji): Photos taken on days 1, 3, and 7 will be processed to calculate the surface area of ecchymosis.

Manual arm circumference measurements: Measurements will be taken with a tape measure to monitor local swelling/inflammation.

Ethical Considerations:

Informed Consent: Participants will be provided with detailed information about the study and will be required to provide informed consent prior to participation.

IRB Approval: The trial will be conducted in compliance with ethical standards and will be reviewed and approved by an Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 undergoing elective arm liposuction.
* No known allergies to TXA or lidocaine.
* BMI < 30.

Exclusion Criteria:

* Previous surgery or trauma to the arms.
* Known coagulation disorders.
* History of thromboembolic events.
* ASA > II.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Ecchymosis of the arms | One week
  NAME OF THE MEASUREMENT: Area of ecchymosis of each arm MEASUREMENT TOOL: Photomicrographic analysis with ImageJ (Fiji) Software. UNIT OF MEASURE: Area (in cm^2) affected by bruising normalized to the total area of the arm (in cm^2).
  Timing: Repeated measures in a standard position and lighting conditions after liposuction on days 1, 3 and 7 postoperatively.

SECONDARY OUTCOMES:
Inflammation of the arm | one week
  NAME OF THE MEASUREMENT: Inflammation of the arms MEASUREMENT TOOL: Metric tape to assess the circumference of the arm. UNIT OF MEASURE: Circumference (in cm) measured at the midpoint of the arm. Timing: Repeated measures in a standard position (90 degree elbow flexion and 90 degree shoulder abduction) after liposuction on days 1, 3 and 7 postoperatively.
Satisfaction | 6 months
  NAME OF THE MEASUREMENT: Aesthetic assessment after liposuction.
  MEASUREMENT TOOL: Global Aesthetic Improvement Scale (GAIS), is a standardized scale used primarily in cosmetic and dermatological treatments to assess the overall aesthetic improvement of a patient after a procedure. It consist of three questions:
  * how do you feel about your appearance after surgery? Possible answers: Very much improved, much improved, slightly improved, no change.
  * Are you satisfied with the surgery? Very satisfied, satisfied, not satisfied.
  * Would you recommend the surgical procedure? Possible answers: Yes, perhaps, no.
  UNIT OF MEASURE: Rate of satisfaction, appearance and recommendation of the procedure.
  Timing: Six months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio E Perez Pachon, MD, Study Director — Department of Plastic Surgery | Scientific Division | Total Definer; Alfredo E Hoyos, MD, Principal Investigator — Department of Plastic Surgery | Total Definer
Locations (1):
- Clinica Dhara, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Our data contains information about highly influential people who are not willing to publicly share their data.

REFERENCES:
- [Background] Wolf Y, Skorochod R, Kwartin S, Shapira L. Tranexamic Acid Irrigation in Liposuction: A Double-Blind, Half-Body, Randomized, Placebo-Controlled Trial. Aesthetic Plast Surg. 2023 Dec;47(6):2525-2532. doi: 10.1007/s00266-023-03499-5. Epub 2023 Jul 24. PMID 37488309
- [Background] Reinhardt ME, Mutyala S, Gerald M, Zhao H, Nova V, Araya Cambronero S, Patel S, Baltodano PA. The Critical Blood-Sparing Effect of Tranexamic Acid (TXA) in Liposuction: A Systematic Review and Meta-Analysis. JPRAS Open. 2023 Feb 2;40:48-58. doi: 10.1016/j.jpra.2023.01.002. eCollection 2024 Jun. PMID 38425698
- [Background] Bayter-Marin JE, Hoyos A, Cardenas-Camarena L, Pena-Pinzon W, Bayter-Torres AF, Diaz-Diaz CA, McCormick-Mendez M, Plata-Rueda EL, Nino-Carreno CS. Effectiveness of Tranexamic Acid in the Postoperative Period in Body Contour Surgery: Randomized Clinical Trial. Plast Reconstr Surg Glob Open. 2023 Nov 15;11(11):e5403. doi: 10.1097/GOX.0000000000005403. eCollection 2023 Nov. PMID 38025645
- [Background] Hoyos AE, Duran H, Cardenas-Camarena L, Bayter JE, Cala L, Perez M, Lopez A, Talleri G, Dominguez-Millan R, Mogollon IR. Use of Tranexamic Acid in Liposculpture: A Double-Blind, Multicenter, Randomized Clinical Trial. Plast Reconstr Surg. 2022 Sep 1;150(3):569-577. doi: 10.1097/PRS.0000000000009434. Epub 2022 Jun 28. PMID 35759637